CLINICAL TRIAL: NCT05434078
Title: Orthofeet: A Prospective Proof of Concept Trial to Evaluate Efficacy, Acceptability, and Perception of Benefit of an Innovative Pain Relief Footwear
Brief Title: Orthofeet: A Prospective Proof of Concept Trial to Evaluate an Innovative Pain Relief Footwear
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bijan Najafi, PhD (Other)
Collaborators: Orthofeet, Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Bijan Najafi, PhD, Principal Investigator, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 51229
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Foot Pain
Keywords: foot pain; falls; frailty; footwear; mobility
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group AB (Active Comparator): Group AB will be started with 6-week Intervention A (OrthoFeet) and then switched to 6-week intervention B (own shoes)
  Interventions: Device: Orthofeet Shoes
- Group BA (No Intervention): Group BA will be started with B (own shoes) for 6 weeks and then switched to Intervention A (OrthoFeet) for the same duration

INTERVENTIONS:
Device: Orthofeet Shoes — Participants will wear a pair of Orthofeet shoes to wear for 6 weeks
  Arms: Group AB

SUMMARY:
The purpose of this prospective randomized crossover study is to evaluate the effectiveness of a new pain relief footwear, Orthofeet, in reducing foot pain and improving daily physical activity. The investigators hypothesize that wearing Orthofeet shoes will lead to a reduction in foot pain, resulting in increased daily physical activity, objectively measured using validated wearable devices.

DETAILED DESCRIPTION:
A clinical study at Baylor College of Medicine is being conducted to evaluate the short- and intermediate-term benefits and effectiveness of a novel pain relief footwear, Orthofeet. This 12-week randomized crossover trial aims to recruit 50 eligible ambulatory adults (aged 50 years or older) with moderate self-reported foot pain. Participants will be randomly assigned to Group AB (25 subjects) or Group BA (25 subjects), with no differences in assessments or eligibility criteria between the groups. In Group AB, participants will wear Orthofeet shoes for 6 weeks, followed by their own shoes for another 6 weeks, while Group BA will follow the reverse order. Pain and function, the primary outcomes, will be measured using the Foot Function Index (FFI), and acceptability will be assessed using a Technology Acceptance Model (TAM) questionnaire. Data will be collected at baseline, 6 weeks, and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older
* self reported foot pain including heel, arch, or ball of foot

Exclusion Criteria:

* Plantar ulcer Patients with major foot deformity (e.g., Charcot foot, Pes Cavus)
* Lower extremity amputation including minor amputation. Foot pain because of nail disorder or keratotic lesions (e.g. corns, calluses)
* unstable conditions such as recent stroke, anticipated changes in medication regime
* Acute fractures of the foot
* Non-ambulatory or unable to stand without help or walk a distance of at least 6 feet without assistance.
* major cognitive impairment or major depression

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Only de-identified data and associated results will be published in peer-reviewed papers or scientific abstracts

REFERENCES:
- [Background] Finco MG, Ouattas A, El-Refaei N, Momin AS, Azarian M, Najafi B. Assessing the Acceptability and Effectiveness of a Novel Therapeutic Footwear in Reducing Foot Pain and Improving Function among Older Adults: A Crossover Randomized Controlled Trial. Gerontology. 2024;70(8):842-854. doi: 10.1159/000539307. Epub 2024 May 22. PMID 38776890
- [Background] Ouattas A, Finco MG, Dehghan Rouzi M, Azarian M, Rojas AZ, Bargas Ochoa M, El-Refaei N, Momin A, Najafi B. The role of therapeutic footwear to increase daily physical activity in older adults with chronic foot pain. Clin Biomech (Bristol). 2025 Mar;123:106373. doi: 10.1016/j.clinbiomech.2024.106373. Epub 2024 Oct 29. PMID 39954566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Baylor Outpatient Clinic (Houston, Texas, USA) via electronic health records, peer referrals, study flyers, and from among participants in prior clinical studies who had agreed to be contacted for new studies. This trial's timeline started at the initial recruitment date of of the firts participant on July 18th, 2022, and concluded at the final follow-up date of August 30th, 2023
Groups:
- OrthoFeet Shoes First, Then Own Shoes: In the group AB (OrthoFeet Shoes first, then Own Shoes), participants wore OrthoFeet shoes for 6 weeks and then their own shoes for another 6 weeks
- Own Shoes First, Then OrthoFeet Shoes: Group BA (Own Shoes first, then OrthoFeet Shoes) followed the reverse order of Group AB, meaning they first wore their own shoes for 6 weeks and then switched to Orthofeet shoes for the subsequent 6 weeks.
Period: Overall Study
Arm/Group | OrthoFeet Shoes First, Then Own Shoes | Own Shoes First, Then OrthoFeet Shoes
Started | 25 | 25
Completed | 22 | 24
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Few subjects were lost to follow up.
Groups:
- OrthoFeet Shoes First, Then Own Shoes: Group AB (OrthoFeet Shoes first, then Own Shoes) started with 6-week Intervention A (OrthoFeet) and then switched to 6-week intervention B (own shoes)
- Own Shoes First, Then OrthoFeet Shoes: Group BA (Own Shoes first, then OrthoFeet Shoes) started with B (own shoes) for 6 weeks and then switched to Intervention A (OrthoFeet) for the same duration
- Total: Total of all reporting groups
Arm/Group | OrthoFeet Shoes First, Then Own Shoes | Own Shoes First, Then OrthoFeet Shoes | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (5) | 66 (5) | 65 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 20 | 23 | 43
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 24 | 46
History of fall [Count of Participants; unit: Participants] | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Foot Pain at Its Worst at Baseline and Week 6
Description: Changes in foot pain from baseline to 6 weeks for each intervention (Orthofeet and own shoes) will be assessed using the Foot Function Index (FFI) questionnaire. The FFI consists of four overall scores, including three subscales: 1) Pain Score (the primary outcome in this study), 2) Disability Score, 3) Activity Limitation Score, and 4) Overall Score.
  The Pain subscale asks participants to rate their foot pain on a scale of 0 (no pain) to 10 (worst imaginable pain), based on their experiences during various activities over the past two weeks. For this outcome, we focused on the FFI pain subscore related to the worst foot pain experienced over the last two weeks.
  To report the final results, participants from intervention A (Orthofeet) and intervention B (own shoes) were combined from groups AB and BA.
Time Frame: baseline, week 6
Population: This study uses a crossover design. Please note that Intervention A comprises data from the first six weeks of Group AB and the last six weeks of Group BA, while Intervention B comprises data from the last six weeks of Group AB and the first six weeks of Group BA. Consequently, the total number of participants is the sum of Group AB and Group BA, which is identical for both Intervention A and Intervention B. Four subjects (out of 50) were lost in follow-up
Measure: Mean (Standard Deviation); unit: unit on scale
Groups:
- OrthoFeet Shoes: Intervention A (OrthoFeet Shoes) involves wearing a pair of OrthoFeet shoes (OrthoFeet©, NJ, USA) for six weeks.
- Own Shoes: Intervention B (Own Shoes, as comparator) involves wearing the participant's own regular shoes for a duration of six weeks.
Arm/Group | OrthoFeet Shoes | Own Shoes
Number analyzed (Participants) | 46 | 46
unit on scale
  Baseline | 6.4 (2.7) | 5.3 (3.2)
  week 6 | 3.6 (2.8) | 5.4 (2.9)

2. Secondary Outcome: Step Count
Description: Step count will be measured over the course of 6 weeks for each intervention arm (Intervention A (Orthofeet) and Intervention B (own shoes)) using a smartwatch (Vivosmart 4, Garmin, USA). Steps per day were recorded in 15-min intervals and summed over each 24-h period. For analysis, the mean daily steps from the last seven consecutive days of each footwear condition (A and B) were calculated for each participant.
Time Frame: from baseline to 6 weeks
Population: Data from twenty-nine participants (out of 46 recruited) with valid physical activity monitoring during both sequences-A (Orthofeet shoes) and B (own shoes)-were included in this secondary analysis. Data from the remaining participants were excluded due to invalid physical activity records.
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | OrthoFeet Shoes | Own Shoes
Number analyzed (Participants) | 29 | 29
steps/day | 5456 (476) | 4758 (474)

3. Secondary Outcome: Daily Energy Expenditure
Description: Active kilocalories (calories burned through physical activity, excluding basal metabolic rate) measured by the smartwatch (Vivosmart watch, Garmin) over the last seven consecutive days were extracted for each intervention period: A (Orthofeet) and B (own shoes). The 90th percentile of daily active kilocalories recorded by the smartwatch from baseline to 6 weeks was included in the analysis.
Time Frame: from baseline to 6 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kcal/day
Arm/Group | Orthofeet Shoes | Own Shoes
Number analyzed (Participants) | 29 | 29
Kcal/day | 532 (119) | 354 (56)

4. Secondary Outcome: Pain Score at Baseline and Week 6
Description: Foot pain at baseline and 6 weeks for each intervention (Orthofeet and own shoes) will be assessed using the Foot Function Index (FFI) questionnaire. The pain subscale asks participants to rate their foot pain on a scale from 0 (no pain) to 10 (worst imaginable pain) based on their experiences during various activities over the past two weeks. Seven of the nine questions were summed for final analysis, excluding "pain walking with orthotics" and "pain standing with orthotics," as the focus was to compare Orthofeet shoes to participants' own shoes, not prescribed orthoses. The resulting total score ranges from 0 to 70, with higher values indicating worse overall pain.
Time Frame: baseline, week 6
Measure: Mean (Standard Deviation); unit: unit on scale
Groups:
- OrthoFeet Shoes: Intervention A (OrthoFeet shoes ) involves wearing a pair of OrthoFeet shoes (OrthoFeet©, NJ, USA) for six weeks.
Arm/Group | OrthoFeet Shoes | Own Shoes
Number analyzed (Participants) | 46 | 46
unit on scale
  baseline | 34.7 (15.9) | 33 (17.5)
  week 6 | 22.8 (16.4) | 31.4 (22.2)

5. Secondary Outcome: Disability at Baseline and Week 6
Description: The disability level at baseline and week 6 was assessed using the disability subscale of the Foot Function Index (FFI). This subscale consists of nine items that evaluate the difficulty experienced in performing various functional activities due to foot problems. These activities include walking inside and outside the house, climbing and descending stairs, getting out of a chair, standing on tiptoe, climbing curbs, and running or fast walking.
  Each item is rated on a scale from 0 (no difficulty) to 10 (so difficult it requires help). The scores for the disability subscale range from 0 to 90, with higher scores indicating greater disability.
Time Frame: baseline, week 6
Measure: Mean (Standard Deviation); unit: unit on scale
Arm/Group | OrthoFeet Shoes | Own Shoes
Number analyzed (Participants) | 46 | 46
unit on scale
  baseline | 38.5 (22.4) | 35.5 (25.5)
  week 6 | 24.9 (8.5) | 31.4 (22.2)

6. Secondary Outcome: Physical Activity Limitation
Description: Physical activity limitations at baseline and were assessed using the Activity Limitation subscale of the Foot Function Index (FFI). This subscale comprises five items that evaluate the extent to which foot problems restrict a person's physical activities, including walking distances, standing on tiptoe, climbing stairs, and engaging in vigorous activities.
  Each item is rated on a scale from 0 (no limitation) to 10 (maximum limitation), with higher scores indicating greater activity limitation. The total score for this subscale ranges from 0 to 50.
  In this study, changes from baseline at week 6 for each intervention duration were assessed and reported.
  In this study the changes from baseline at week 6 for each intervention duration was assessed and reported
Time Frame: baseline, week 6
Measure: Mean (Standard Deviation); unit: unit on scale
Arm/Group | Orthofeet Shoes | Own Shoes
Number analyzed (Participants) | 46 | 46
unit on scale
  baseline | 13.3 (9.4) | 12.2 (10)
  week 6 | 9.9 (8.5) | 10.5 (8.7)

7. Secondary Outcome: Daily Metabolic Equivalent of Task (METS)
Description: We used a Garmin smartwatch to report the Daily Metabolic Equivalent of Task (METs). Median daily MET values over the last seven consecutive days for each participant, during each footwear condition (Orthofeet shoes and their own shoes), were calculated following the guidelines of the American College of Sports Medicine (ACSM) and the American Heart Association (AHA) (Haskell et al., 2007).
  To calculate MET-minutes per week (MET·min·wk-¹), the median daily METs were multiplied by 60, as recommended by ACSM and AHA. The mean values for the calculated "Median daily MET" across all participants, during periods when they wore Orthofeet shoes and their own shoes, were computed and reported.
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: MET-minutes per week
Arm/Group | OrthoFeet Shoes | Own Shoes
Number analyzed (Participants) | 29 | 29
MET-minutes per week | 461 (22) | 427 (17)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: An adverse event (AE) is any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (e.g., worsening foot pain, falls, allergy), symptom, or disease, temporally associated with the participant's involvement in the research, whether or not considered related to their participation.
Arm/Group | Orthofeet Shoes | Own Shoes
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 0/46 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT05434078/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/78/NCT05434078/ICF_001.pdf